CLINICAL TRIAL: NCT06812741
Title: Comparison of Mean Duration of Postoperative Analgesia in Patients Undergoing Inguinal Hernia Surgery Treated with Transversus Abdominal Plane Block Vs Ilioinguinal and Iliohypogastric Nerve Blocks
Brief Title: Duration of Postop Analgesia After Inguinal Hernia Surgery Treated with TAP Block Vs II/IH Nerve Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pakistan Navy Station Shifa Hospital (Other)
Responsible Party: Principal Investigator, Kenan Anwar Khan, FCPS Registrar in Anaesthesia, Pakistan Navy Station Shifa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 530/ 2024
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Analgesia
Keywords: postop analgesia; postoperative analgesia; TAP block; transversus abdominis plane block; ilioinguinal/ iliohypogastric nerve block; ilioinguinal/iliohypogastric nerve block; inguinal hernia surgery; abdominal nerve block; nerve block; nerve blocks; bupivacaine; ultrasound guided nerve block; ultrasound guided nerve blocks; 0.25% bupivacaine; 0.25 percent bupivacaine; hernioplasty; internal oblique; transversus abdominis; IIN; IHN; IIN/ IHN; II/ IH nerve block; transversus abdominis muscle; ilioinguinal muscle; iliohypogastric muscle
MeSH Terms: interventions — Dental Occlusion; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inguinal Hernia Surgery (Group T) (Experimental): Half of the study participants named Group T were administered Ultrasound Guided Transversus Abdominis Plane Nerve Block and the other half named Group I were administered Ilioinguinal & Iliohypogastric Nerve Block before the Inguinal Hernia Surgery.
  Interventions: Drug: Transversus abdominis plane (TAP) block with 0.25 % bupivacaine
- Inguinal Hernia Surgery (Group I) (Experimental): Half of the study participants named Group T were administered Ultrasound Guided Transversus Abdominis Plane Nerve Block and the other half named Group I were administered Ilioinguinal & Iliohypogastric Nerve Block before the Inguinal Hernia Surgery.
  Interventions: Drug: Ilioinguinal/iliohypogastric Nerve Block with 0.25 % bupivacaine

INTERVENTIONS:
Drug: Transversus abdominis plane (TAP) block with 0.25 % bupivacaine — The probe was placed in a plane transverse to the lateral abdominal wall in the mid-axillary line immediately cephalad to the iliac crest. The needle was advanced immediately anterior to the probe using the in-plane needle-probe orientation and advanced posteriorly until the needle was observed to penetrate the interface between the internal oblique and transversus abdominis muscles. Thereafter, a local anesthetic (0.2 mL/kg of 0.25 % bupivacaine) was injected incrementally, and the spread was observed within the plane.
  Arms: Inguinal Hernia Surgery (Group T)
Drug: Ilioinguinal/iliohypogastric Nerve Block with 0.25 % bupivacaine — The ultrasound probe was placed immediately medial and slightly cephalad to the upper aspect of the anterior superior iliac spine to obtain a short-axis view of the nerves situated between the two abdominal muscles (internal oblique and transversus abdominis), A 22 G needle tip ~1 cm caudal to the probe surface was introduced and was advanced until a characteristic 'tenting' of the interface between the two muscles was seen and was then further advanced deep to this interface until a pop was felt and then the injectate (0.2 mL/kg of 0.25 % bupivacaine) was observed spreading between these two layers.
  Arms: Inguinal Hernia Surgery (Group I)

SUMMARY:
Comparing Postop Analgesia after Inguinal Hernia Surgery treated with TAP Block Vs Ilioinguinal/ Iliohypogastric Nerve Block

DETAILED DESCRIPTION:
Comparison of Mean Duration of Postoperative Analgesia in Patients undergoing Inguinal Hernia Surgery treated with Transversus Abdominal Plane Block Versus Ilioinguinal/ Iliohypogastric Nerve Block

ELIGIBILITY:
Inclusion Criteria:

* Patients giving written informed consent
* Patients undergoing Inguinal Hernia surgery
* patients with ages 18-60 years
* ASA 1 and 2 patients

Exclusion Criteria:

* INR > 1.0 (patients with bleeding tendency)
* EF < 45 % (patients with cardiac dysfunction)
* FEV1 < 80 % of normal (patients with pulmonary dysfunction)
* patients with renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Mean duration of Postoperative Analgesia | 6 months
  The study was conducted to compare the mean duration of postoperative analgesia in patients undergoing inguinal hernia repair surgery treated with transversus abdominis plane block versus the mean duration of postoperative analgesia in patients undergoing inguinal hernia repair surgery treated with ilioinguinal and iliohypogastric nerve block.

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Military Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No